CLINICAL TRIAL: NCT05590468
Title: Randomized, Double-blinded, Placebo-controlled Study Evaluating the Efficacy of Nicotinamide Riboside (NR) - a Vitamin B3 Derivative - for Treatment of Mitochondrial Myopathy Disorder
Brief Title: A Study to Evaluate Vitamin B3 Derivative to Treat Mitochondrial Myopathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ralitza Gavrilova (Other)
Responsible Party: Sponsor-Investigator, Ralitza Gavrilova, Regulatory Sponsor, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-005125
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Mitochondrial Myopathy
MeSH Terms: conditions — Mitochondrial Myopathies | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotinamide Riboside treatment group (Experimental): Subjects will receive vitamin B3 derivative Nicotinamide Riboside (NR) daily for 12 months
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo Group (Placebo Comparator): Subjects will receive a placebo daily for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Vitamin B3 derivative; a total of 1000 mg/day in a regimen of 500mg every 12 hours by mouth (either fasting or fed)
  Arms: Nicotinamide Riboside treatment group
Drug: Placebo — Looks exactly like the study drug, but it contains no active ingredient
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to determine the effects of Nicotinamide Riboside (NR) supplement in adult-onset symptoms of mitochondrial myopathy.

ELIGIBILITY:
Inclusion Criteria:

* Biochemically and/or genetically confirmed or confirmed primary mitochondrial myopathy based on published diagnostic criteria.
* Biochemically confirmed mitochondrial disorder would mean that the patient meets clinical criteria and has either biopsy or biochemical testing that supports the diagnosis.
* Confirmed mitochondrial disorder means that the patient meets published clinical criteria for the diagnosis and has also had confirmatory genetic testing for the disorder type.
* Agreed to avoid vitamin supplementation or nutritional products with vitamin B3 forms 14 days prior to the enrollment and during the study in order to not exceed 200 mg/day of vitamin B3 derivatives intake.
* Female of childbearing potential agreed to use effective contraception throughout the study.
* Written, informed consent to participate in the study.

Exclusion Criteria:

* Unwilling to comply with the follow-up schedule.
* Inability or refusal to give informed consent by the patient or a legally authorized representative.
* Known pregnancy or breastfeeding.
* Concurrent participation in another investigational drug study or within washout period of treatment.
* Presence of other medical symptoms or condition, which may interfere with interpretation of outcome measures as determined by the study PI.

Clinical / Laboratory Exclusion Criteria:

* Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min.
* Patients in permanent Renal Replacement Therapy.
* Serum alkaline phosphatase 50% above normal limit.
* Serum aspartate transaminase 50% above normal limit.
* Serum Thyroxine (T4) 50% above or below normal limit.
* Serum Thyroid Stimulating Hormone (TSH) 50% above or below normal limit.
* Severe anemia with Hb < 7g/dL.
* Severe leukocytosis with WBC > 15,000/mm^3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Changes in 6-Minute Walk Test Performance | Baseline, 6 months, 12 months
  The 6-minute walk test (6MWT) quantifies the distance a person can walk in six minutes. Measured in meters.

SECONDARY OUTCOMES:
Change in skeletal muscle function | Baseline, 6 months, 12 months
  Measured using the Short Physical Performance Battery (SPPB) score based on timed measures of standing balance, walking speed and ability to rise from a chair. Each of the 3 performance measures will be assigned a score ranging from 0 to 4, with 4 indicating the highest level of performance and 0 the inability to complete the test. A summary score (range 0-12) will be subsequently calculated by adding the 3 scores.
Change in skeletal muscle strength | Baseline, 6 months, 12 months
  Measured using the strength one repetition maximum (1RM leg press) defined as the maximal weight an individual can lift for only one repetition with correct technique.
Change in isometric strength of trunk flexors | Baseline, 6 months, 12 months
  Assessed by generated maximum force against a stationary dynamometer reported in kilograms of force. Trunk flexion strength tested in the supine position with knees slightly bent, arms at side and head in midline. The base of the dynamometer will be placed on the middle of the sternum and the patient will be instructed to exert isometric force by lifting both scapula off the plinth.
Change in isometric strength of trunk extensor muscle | Baseline, 6 months, 12 months
  Assessed by generated maximum force against a stationary dynamometer reported in kilograms of force. Trunk extensor muscle strength tested in prone position. The base of the dynamometer will be placed at the level of the T4 spine and the patient instructed to generate an isometric force by lifting the chest off the plinth. After sufficient practice in the standardized positions, 5 trials will be recorded in each position.
Change in maximal oxygen uptake (VO2 max) | Baseline, 6 months, 12 months
  Maximal oxygen uptake (VO2 max) test measures the maximum rate of oxygen consumption during incremental exercise (exercise of increasing intensity) and reflects the cardiorespiratory fitness of an individual. Reported in ml/kg/min.

CONTACTS AND LOCATIONS:
Overall Officials: Ralitza H. Gavrilova, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No